CLINICAL TRIAL: NCT06166797
Title: Elucidating Growth Hormone Dynamics at Stages of Progressive Nonalcoholic Fatty Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Takara Stanley, Associate Professor of Pediatrics, Massachusetts General Hospital
Other Study IDs: 2021p-003599
Record Dates: First submitted 2023-11-17; First posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- No NAFLD: individuals with <5 percent hepatic fat fraction on magnetic resonance spectroscopy
- Simple Steatosis: individuals with at least 10% fat fraction on magnetic resonance spectroscopy without any history of nonalcoholic steatohepatitis or evidence of fibrosis
- Nonalcoholic Steatohepatitis: individuals with biopsy confirmed nonalcoholic steatohepatitis and stage 2 or 3 fibrosis

SUMMARY:
The purpose of this study is to investigate relationships between the body's growth hormone "axis" and nonalcoholic fatty liver disease. The growth hormone "axis" includes the hormones growth hormone and insulin-like growth factor 1, and associated proteins. We hypothesize that there will be a relationship such that people with more advanced nonalcoholic fatty liver disease will have greater impairments in the growth hormone axis. There are no treatments associated with this research study.

DETAILED DESCRIPTION:
Several lines of existing research implicate activity of the GH/IGF-1 axis in the development of nonalcoholic fatty liver disease (NAFLD) and nonalcoholic steatohepatitis (NASH) in humans. Careful phenotyping of GH dynamics in individuals with NAFLD and NASH is required for comprehensive understanding of the degree to which perturbations in the GH axis contribute to the pathogenesis of NAFLD/NASH. The purpose of this research is to comprehensively assess GH dynamics in individuals across the spectrum of NAFLD to determine associations between the GH/IGF-1 axis and stages of disease progression in NAFLD.

ELIGIBILITY:
Inclusion criteria:

Men 18-70yo

* BMI between 25kg/m2 - 40kg/m2.
* Hepatitis C antibody and Hepatitis B surface antigen negative.
* Meet inclusion criteria for one of Groups 1-3 based on medical history, laboratory criteria, and hepatic fat fraction (1H-MRS) and/or liver biopsy

  * Group 1: No NAFLD: no history of NAFLD/NASH, hepatic fat fraction <5% on 1H-MRS, ALT < 30 U/L.
  * Group 2: Simple Steatosis: no history of NASH, hepatic fat fraction ≥10% on 1H-MRS, ALT < 30 U/L.
  * Group 3: Nonalcoholic Steatohepatitis: Biopsy confirmed NASH within the year prior to study participation, with liver fibrosis stage 2 or 3 on biopsy.

Exclusion criteria:

* Heavy alcohol use defined as consumption of > 30mg daily for at least 3 consecutive months over the past 5 years
* Type 1 diabetes, any use of insulin, or any use of other anti-diabetes medication except metformin or sulfonylurea. Individuals with Type 2 diabetes that is controlled by diet or by metformin and/or sulfonylurea will be eligible.
* Use of any specific pharmacological treatments for NAFLD/NASH except vitamin E within the 3 months before screening visit.
* Chronic systemic corticosteroid use in the ≤6 months prior to the baseline visit.
* Chronic use of Actigall, methotrexate, amiodarone, or tamoxifen
* Known diagnosis of alpha-1 antitrypsin deficiency, Wilson's disease, hemochromatosis, or autoimmune hepatitis
* Use of GH or GHRH within the past 6 months
* Change in lipid lowering or anti-hypertensive regimen within 2 months of screening
* Hemoglobin < 12.5 g/dL
* Severe chronic illness judged by the investigator to present a contraindication to participation
* History of hypopituitarism, head irradiation or any other condition known to affect the GH axis.
* Use of testosterone or estrogen or progesterone unless physiologic stable testosterone use for at least 1 year prior to study entry
* Routine MRI exclusion criteria such as the presence of a pacemaker or cerebral aneurysm clip
* Weight loss surgery within 1 year before baseline. Weight loss surgery more than 1 year prior to baseline visit is permissible if no active weight loss (<10% decrease in weight over past 6 months)
* Lack of fluency in English and/or inability to complete the consent process in English.
* Judge by the investigator to be inappropriate for the study for other reasons not detailed above.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Men 18-70yo with or without nonalcoholic fatty liver disease
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
peak growth hormone | at baseline
  peak growth hormone level during standard 3-hour glucagon stimulation test

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital; Takara Stanley, MD, Principal Investigator — Massachusetts General Hospital

IPD SHARING:
Plan to Share IPD: Undecided